CLINICAL TRIAL: NCT00821444
Title: Phase 1 Study Of Ziprasidone Pharmacokinetics Of Reduced Food Effect Formulation B16 Under Fed And Fasting Conditions Compared To Commercial Geodon Capsules Under Fed Conditions In Healthy Subjects
Brief Title: Ziprasidone Pharmacokinetics Using a Reduced Food Effect Formulation Compared to Pharmacokinetics From Commercial Capsules
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A1281191
Record Dates: First submitted 2009-01-09; First posted 2009-01-13 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Healthy
Keywords: schizophrenia, pharmacokinetics, bioavailability, food effect
MeSH Terms: conditions — Schizophrenia | interventions — ziprasidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Geodon fed (Active Comparator): Commercial Geodon (ziprasidone) capsules given with food
  Interventions: Drug: ziprasidone
- B16 Fasted (Experimental): Experimental reduced food effect formulation given without food
  Interventions: Drug: B16 Fasted
- B16 Fed (Experimental): Experimental reduced food effect formulation given with food
  Interventions: Drug: B16 Fed

INTERVENTIONS:
Drug: ziprasidone — 40 mg capsule, single dose x 3
  Other Names: Geodon, Zeldox
  Arms: Geodon fed
Drug: B16 Fasted — 40 mg tablet, single dose X 3
  Arms: B16 Fasted
Drug: B16 Fed — 40 mg tablet, single dose X 3
  Arms: B16 Fed

SUMMARY:
Commercial ziprasidone capsules show a large increase in bioavailability with food. The formulation tested in this study aims to reduce or eliminate that increase.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects
* Signed informed consent document

Exclusion Criteria:

* Any significant physical or psychological disease
* Concomitant administration of other pharmaceuticals

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2009-01; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Relative bioavailability measured as geometric mean ratios of AUCinf and Cmax and the associated 90% confidence intervals calculated for various pairs of study treatments. | 2 months

SECONDARY OUTCOMES:
Adverse events reported, laboratory test results, vital signs observed with each study treatment | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1281191&StudyName=Ziprasidone%20pharmacokinetics%20using%20a%20reduced%20food%20effect%20formulation%20compared%20to%20pharmacokinetics%20from%20commercial%20capsules